CLINICAL TRIAL: NCT02809404
Title: Dried Blood SPOT Analysis of Everolimus in Cancer Patients
Brief Title: Dried Blood SPOT Analysis of Everolimus in Cancer Patients (SPOT-study)
Acronym: SPOT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MOMAM15-SPOT
Record Dates: First submitted 2016-06-01; First posted 2016-06-22 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2016-05

CONDITIONS: Breast Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and drop of blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Everolimus
  Other Names: Afinitor

SUMMARY:
Everolimus shows a large interpatient variability with fixed dose administration. These very different exposure levels between individuals can result in supratherapeutic or subtherapeutic exposure levels and consequently in over- or undertreatment, respectively. Dose individualization based on the measured drug concentration could theoretically result in less toxicity and more efficacy.

Nowadays everolimus exposure is determined by everolimus concentration in whole blood. Therefore, a vena puncture is always necessary. This is invasive and requires patients to come to the hospital. It would be convenient for patients to have their everolimus blood concentration determined by dried blood spot (DBS) analysis. With DBS only a single drop of blood from the finger is necessary, which can be done at home and sent by regular mail for analysis. Previous studies have shown the feasibility of this approach. In patients with cancer treated with everolimus 10mg once daily, the correlation between everolimus DBS concentrations and whole blood concentration is yet unknown. Therefore, the investigators want to determine the everolimus concentration collected with DBS from a finger prick with everolimus concentration from whole blood and everolimus concentration collected with DBS from whole blood.

In addition, possibly a relatively high everolimus concentration in saliva could be correlated with the incidence and severity of oral mucositis. Determination of drug concentration in saliva has also been proven to be feasible before.

Therefore, in this study the investigators want to determine whether the everolimus concentration in saliva correlates with the incidence of oral mucositis and how everolimus concentration in saliva correlates with everolimus concentration in whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently treated with everolimus for any type of cancer
* Patients from whom it is possible to collect blood samples
* At least 18 years of age
* Able and willing to sign the Informed Consent Form prior to study assessments.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently treated with everolimus for any type of cancer are eligible in this study.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlation everolimus concentration DBS with whole blood | Up to 2 years
  Correlation between trough everolimus concentration from DBS analysis collected with finger prick with trough everolimus concentration in whole blood, measured at any time during everolimus treatment

SECONDARY OUTCOMES:
Correlation everolimus concentration whole blood with saliva | Up to 2 years
  Correlation between trough everolimus concentration from whole blood with trough everolimus concentration in saliva, measured at any time during everolimus treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nielka van Erp, PharmD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands